CLINICAL TRIAL: NCT02273739
Title: A Phase 1/2, Multicenter, Open-Label, Dose-Escalation Study of AG-221 in Subjects With Advanced Solid Tumors, Including Glioma, and With Angioimmunoblastic T-cell Lymphoma, That Harbor an IDH2 Mutation
Brief Title: Study of Orally Administered Enasidenib (AG-221) in Adults With Advanced Solid Tumors, Including Glioma, or Angioimmunoblastic T-cell Lymphoma, With an IDH2 Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AG221-C-003; 2014-003424-47 (EudraCT Number)
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2014-10-16; First posted 2014-10-24 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Solid Tumor; Glioma; Angioimmunoblastic T-cell Lymphoma; Intrahepatic Cholangiocarcinoma; Chondrosarcoma
Keywords: solid tumor; intrahepatic cholangiocarcinoma; chondrosarcoma; angioimmunoblastic T-cell lymphoma; AITL; IDH; glioma; solid tumor, including intrahepatic cholangiocarcinoma and chondrosarcoma
MeSH Terms: conditions — Glioma; Immunoblastic Lymphadenopathy; Cholangiocarcinoma; Chondrosarcoma | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enasidenib (Experimental): During the dose escalation phase, consented eligible participants will be enrolled into sequential cohorts of increasing doses of enasidenib.The starting dose for this study is 100 mg administered every 24 hours,
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Enasidenib tablets administered orally once a day in 28-day treatment cycles until disease progression or unacceptable toxicities.
  Other Names: AG-221; IDHIFA®

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and clinical activity of enasidenib in adults with advanced solid tumors, including glioma, or with angioimmunoblastic T-cell lymphoma (AITL), with an isocitrate dehydrogenase-2 (IDH2) mutation.

DETAILED DESCRIPTION:
The first portion of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of enasidenib to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose. The second portion of the study is a planned dose expansion phase where three cohorts of patients will receive enasidenib to further evaluate the safety, tolerability, and clinical activity. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

Enrollment into the AG221-C-003 study was closed following enrollment of the dose escalation Cohort 4 (650 mg QD) in order to focus resources on the development of other pipeline IDH inhibitors in solid tumors, gliomas, and lymphoma; it was not due to safety reasons. Participants receiving enasidenib at the time of study closure were to be allowed to continue treatment until disease progression or the development of unacceptable toxicity, as outlined in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age
* Histologically or cytologically confirmed advanced solid tumor, including glioma, or angioimmunoblastic T-cell lymphoma (AITL) that has recurred or progressed following standard therapy, or that has not responded to standard therapy
* Subjects must be amenable to peripheral blood sampling, urine sampling, and biopsies during the study. Subjects with AITL must also be amenable to serial bone marrow biopsies
* Documented IDH2 gene-mutated disease based on local site testing
* Measurable disease by RECIST v1.1 for subjects with solid tumors without glioma, by modified RANO criteria for subjects with glioma, or by the revised IWG criteria for subjects with AITL
* Subjects must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Adequate bone marrow function (subjects other than those with AITL) as evidenced by: absolute neutrophil count ≥ 1.0 ×10^9/L; hemoglobin > 9 g/dL (subjects may be transfused red blood cells to this level.); platelets ≥ 50 × 10^9/L
* Adequate hepatic function as evidenced by: serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease, a gene mutation in UGT1A1, or disease involvement, following approval by the Medical Monitor; aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 2.5 × ULN, with the exception of subjects with bone metastases and/or suspected disease-related liver or biliary involvement, where ALP must be ≤ 5 × ULN
* Adequate renal function as evidenced by: serum creatinine ≤ 2.0 × ULN; OR creatinine clearance > 40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
* Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy. Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days (females and males) following the last dose of AG-221
* Previous allogeneic stem cell transplant is allowed only if subjects are >100 days from stem cell transplant and do not have uncontrolled acute or chronic graft-vs-host disease

Exclusion Criteria:

* Received systemic anticancer therapy or radiotherapy < 21 days prior to their first day of study drug administration
* Received an investigational agent < 14 days prior to their first day of study drug administration. In addition, the first dose of AG-221 should not occur before a period ≥ 5 half-lives of the investigational agent has elapsed
* Subjects taking the following sensitive cytochrome P450 (CYP) substrate medications that have a narrow therapeutic range are excluded from the study unless they can be transferred to other medications prior to enrolling: paclitaxel (CYP2C8), warfarin, phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline and tizanidine (CYP1A2)
* Subjects taking the P-glycoprotein (P-gp) and breast cancer resistant protein (BCRP) transporter-sensitive substrates digoxin and rosuvastatin should be excluded from the study, unless they can be transferred to other medications prior to enrolling. study unless they can be transferred to other medications prior to enrolling
* Subjects for whom potentially curative anticancer therapy is available
* Pregnant or breastfeeding
* Active severe infection that required anti-infective therapy or with an unexplained fever > 38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, subjects with tumor fever may be enrolled)
* Known hypersensitivity to any of the components of AG-221
* Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of Cycle 1Day 1
* History of myocardial infarction within the last 6 months
* Subjects with uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg) are excluded. Subjects requiring 2 or more medications to control hypertension are eligible with Medical Monitor approval.
* Known unstable or uncontrolled angina pectoris
* Known history of severe and/or uncontrolled ventricular arrhythmias
* Heart-rate corrected QT (QTc) interval > 450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with right bundle branch block and a prolonged QTc interval should be reviewed by the Medical Monitor for potential inclusion
* Subjects taking medications that are known to prolong the QT interval
* Known infection with human immunodeficiency virus (HIV) or active hepatitis B or C
* Any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Subjects with brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery, or other therapy, including to control symptoms, within 2 months of first dose. Subjects with glioma who are on a stable, steroid-dosing regimen prior to screening magnetic resonance imaging (MRI) may be permitted to enroll with Medical Monitor approval
* In subjects with AITL, evidence of meningeal or cerebral disease or a history of progressive multifocal leukoencephalopathy
* Radiotherapy involving < 25% of the hematopoietically active bone marrow within 21 days preceding first dose of study treatment
* Radiotherapy involving ≥ 25% of the hematopoietically active bone marrow within 42 days preceding first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Agios Pharmaceuticals, Inc.
Locations (11):
- United States (9):
  - Los Angeles, California
  - Miami, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Omaha, Nebraska
  - New York, New York
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Dallas, Texas
- France (2):
  - Bordeaux
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 clinical sites in the United States and France. The study was to include a dose escalation phase to determine maximum tolerated dose (MTD) followed by expansion cohorts to further evaluate the safety and tolerability of the MTD. Enrollment was closed following enrollment of the dose escalation Cohort 4 and the expansion phase was not conducted.
Pre-assignment Details: Participants with advanced solid tumors, including glioma, or angioimmunoblastic T-cell lymphoma (AITL) were enrolled into sequential cohorts of increasing doses of enasidenib in the dose-escalation phase of the study.
Groups:
- Enasidenib 100 mg: Participants received enasidenib 100 mg tablets once a day (QD) on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
- Enasidenib 200 mg: Participants received enasidenib 200 mg tablets QD on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
- Enasidenib 400 mg: Participants received enasidenib 400 mg tablets QD on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
- Enasidenib 650 mg: Participants received enasidenib 650 mg tablets QD on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Started | 3 | 4 | 7 | 7
Completed (Participants ongoing treatment) | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 7 | 7
Not completed — Progression of Disease | 3 | 4 | 5 | 2
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled particpants
Groups:
- Enasidenib 100 mg: Participants received enasidenib 100 mg tablets QD on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg | Total
Number analyzed (Participants) | 3 | 4 | 7 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (16.80) | 68.0 (5.10) | 52.0 (18.47) | 61.3 (13.34) | 58.8 (14.97)
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 1 | 0 | 4 | 3 | 8
  60 to < 70 years | 1 | 3 | 2 | 1 | 7
  70 to < 75 years | 1 | 0 | 1 | 2 | 4
  ≥ 75 years | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 3 | 8
  Male | 2 | 4 | 3 | 4 | 13
Race [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 4 | 6 | 4 | 16
  Not Reported | 0 | 0 | 1 | 3 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subjects disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis.
  * 0 = Fully Active (Most Favorable Activity);
  * 1 = Restricted activity but ambulatory;
  * 2 = Ambulatory but unable to carry out work activities;
  * 3 = Limited Self-Care;
  * 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 1 | 2 | 3 | 3 | 9
    1= Restricted but Ambulatory | 0 | 2 | 2 | 2 | 6
    2 = Ambulatory but Unable to Work | 2 | 0 | 2 | 2 | 6
    3 = Limited Self-Care | 0 | 0 | 0 | 0 | 0
    4 = Completely Disabled | 0 | 0 | 0 | 0 | 0
Tumor Type [Count of Participants; unit: Participants]
  Cholangiocarcinoma | 0 | 0 | 1 | 3 | 4
  Chondrosarcoma | 1 | 1 | 1 | 0 | 3
  Glioma | 1 | 0 | 4 | 1 | 6
  Angioimmunoblastic T-cell lymphoma (AITL) | 1 | 1 | 0 | 3 | 5
  Other | 0 | 2 | 1 | 0 | 3
Isocitrate dehydrogenase 2 (IDH2) Mutation Type [Count of Participants; unit: Participants] — Isocitrate dehydrogenase 2 (IDH2) gene mutations have been described in patients with gliomas, chondrosarcomas, intrahepatic cholangiocarcinomas, as well as a variety of other solid and liquid tumors. Mutations in IDH2 most commonly lead to alterations affecting arginine-172 (R172) or arginine-140 (R140) in IDH2. The mutated protein shows a gain-of-function, neomorphic activity, catalyzing the reduction of alpha-ketoglutarate (α-KG) to 2-hydroxyglutarate (2-HG), an oncogenic metabolite.
  Mutation in IDH2 was required for study entry.
  Participants
    R172 | 3 | 3 | 3 | 6 | 15
    R140 | 0 | 0 | 0 | 0 | 0
    Other | 0 | 1 | 3 | 1 | 5
    Missing | 0 | 0 | 1 | 0 | 1
Isocitrate dehydrogenase (IDH) 1 Gene Result [Count of Participants; unit: Participants] — IDH1 mutations have been found in those with both blood and solid tumors; mutations in IDH1 and IDH2 are almost always mutually exclusive and occur at very early stages of tumor development suggesting that they promote formation and progression of tumors. Mutations in the IDH1 protein most commonly lead to alterations affecting arginine-132 (R132H or R132C)
  Participants
    IDH1 R132 | 0 | 0 | 0 | 0 | 0
    Negative | 2 | 4 | 6 | 4 | 16
    Other | 0 | 0 | 0 | 3 | 3
    Missing | 1 | 0 | 1 | 0 | 2
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] — BSA is the total surface area of the body. BSA was calculated as weight (kilograms)^0.425 x height (cm)^0.725 / 139.2.
  m² | 1.8 (0.21) | 2.1 (0.15) | 1.8 (0.23) | 1.8 (0.18) | 1.8 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events included any adverse events (AEs) occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of the study drug. Severity was graded according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03 or according to the following scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5= Fatal, death related to AE.
  A serious AE is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required or prolonged existing inpatient hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event.
  Relationship to study drug administration was determined by the investigator as not related, possibly related, or probably related; all AEs classified as possibly or probably related were considered treatment-related.
Time Frame: From first dose of study drug to 28 days after last dose; median (minimum, maximum) duration of exposure was 66 (8, 197) days across all cohorts.
Population: All participants who were enrolled and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 7 | 7
Participants
  ≥ 1 treatment-emergent adverse event (TEAE) | 3 | 4 | 6 | 7
  ≥ 1 treatment-related TEAE | 3 | 4 | 5 | 5
  ≥ 1 Grade 3/4 TEAE | 2 | 3 | 5 | 4
  ≥ 1 Grade 3/4 treatment-related TEAE | 0 | 0 | 3 | 3
  ≥ 1 Grade ≥ 3 TEAE | 2 | 3 | 5 | 5
  ≥ 1 Grade ≥ 3 treatment-related TEAE | 0 | 0 | 3 | 3
  ≥ 1 Grade 5 TEAE | 1 | 0 | 1 | 2
  ≥ 1 Grade 5 treatment-related TEAE | 0 | 0 | 0 | 0
  ≥ 1 serious TEAE | 2 | 2 | 3 | 4
  ≥ 1 serious treatment-related TEAE | 0 | 0 | 0 | 2
  ≥ 1 TEAE leading to discontinuation of enasidenib | 0 | 0 | 0 | 3
  ≥ 1 treatment-related TEAE leading to discontinuation of enasidenib | 0 | 0 | 0 | 1
  ≥ 1 TEAE leading to dose reduction of enasidenib | 0 | 0 | 0 | 0
  ≥ 1 treatment-related TEAE leading to dose reduction of enasidenib | 0 | 0 | 0 | 0
  ≥ 1 TEAE leading to interruption of enasidenib | 0 | 2 | 3 | 5
  ≥ 1 treatment-related TEAE leading interruption of enasidenib | 0 | 0 | 2 | 4
  ≥ 1 TEAE leading to death | 1 | 0 | 1 | 2
  ≥ 1 treatment-related TEAE leading to death | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: Toxicities were graded and documented according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03. A dose-limiting toxicity (DLT) was defined as an event considered related to enasidenib and meeting 1 of the following criteria:
  Non-hematologic:
  - All clinically significant non-hematologic toxicities CTCAE ≥ Grade 3, considered not related to underlying disease or intercurrent illness, with the exception of ≥ Grade 3 blood bilirubin increases in participants with a uridine diphosphate-glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) mutation. In participants with a UGT1A1 mutation, blood bilirubin increases of > 5 × upper limit of normal (ULN) were considered a DLT.
  Hematologic:
  - Drug-related, prolonged myelosuppression of ≥ Grade 4 neutropenia or thrombocytopenia lasting beyond Day 28 of Cycle 1 unless related to bone marrow involvement by AITL.
Time Frame: Cycle 1 (28 days)
Population: All enrolled and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 7 | 7
Participants | 0 | 0 | 1 | 0

3. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at Each Visit
Description: ECOG performance status is used by doctors and researchers to assess how a subjects disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis.
  * 0 = Fully active (most favorable activity);
  * 1 = Restricted activity but ambulatory;
  * 2 = Ambulatory but unable to carry out work activities;
  * 3 = Limited self-care;
  * 4 = Completely disabled, no self-care (least favorable activity).
Time Frame: Baseline, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, and at end of treatment
Population: Enrolled participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 7 | 7
score on a scale
  Baseline | 1.3 (1.15) | 0.5 (0.58) | 0.9 (0.90) | 0.9 (0.90)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 4 | 5 | 5
  Cycle 1 Day 15 | 1.7 (0.58) | 1.8 (1.50) | 0.8 (0.84) | 1.0 (0.71)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 5 | 3
  Cycle 2 Day 1 | 1.7 (0.58) | 0.8 (0.50) | 1.2 (1.30) | 0.7 (0.58)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 0 | 2 | 2
  Cycle 3 Day 1 | 1.0 |  | 1.0 (0.00) | 1.0 (0.00)
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 2 | 1
  Cycle 4 Day 1 | 1.0 |  | 1.0 (0.00) | 1.0
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 1
  Cycle 5 Day 1 |  |  | 1.0 (0.00) | 1.0
  End of Treatment: number analyzed (Participants) | 2 | 3 | 4 | 3
  End of Treatment | 2.5 (0.71) | 0.7 (0.58) | 1.3 (1.50) | 1.7 (1.15)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) After a Single Dose of Enasidenib on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for assessment of enasidenib pharmacokinetics (PK).
  Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Enasidenib 100 mg: Participants received a single oral dose of enasidenib 100 mg on Day -3.
- Enasidenib 200 mg: Participants received a single oral dose of enasidenib 200 mg on Day -3.
- Enasidenib 400 mg: Participants received a single oral dose of enasidenib 400 mg on Day -3.
- Enasidenib 650 mg: Participants received a single oral dose of enasidenib 650 mg on Day -3.
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
ng/mL | 1403.4 (77.9) | 1433.0 (51.2) | 4540.6 (63.7) | 4702.9 (61.3)

5. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Enasidenib After a Single Dose on Day -3
Description: as for outcome 4
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
hours | 2.0 [2 to 8] | 6.1 [2 to 25] | 8.0 [2 to 10] | 3.3 [2 to 24]

6. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 10 Hours Postdose (AUC0-10) of Enasidenib After a Single Oral Dose on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for assessment of enasidenib pharmacokinetics (PK).
  Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
h*ng/mL | 10031.7 (79.0) | 11040.2 (55.9) | 31959.0 (56.7) | 29847.8 (59.6)

7. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 72 Hours Postdose (AUC0-72) of Enasidenib After a Single Dose on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3) for assessment of enasidenib pharmacokinetics (PK).
  Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 72 hours post-dose (AUC0-72) was calculated using the linear trapezoidal rule.
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
h*ng/mL | 62420.0 (80.6) | 86900.7 (62.5) | 206214.4 (65.2) | 248315.9 (69.9)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metabolite AGI-16903 After a Single Dose of Enasidenib on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3).
  AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Day -3 pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
ng/mL | 94.2 (64.5) | 71.9 (70.8) | 273.0 (52.9) | 239.4 (64.8)

9. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Metabolite AGI-16903 After a Single Dose of Enasidenib on Day -3
Description: as for outcome 8
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
hours | 70.3 [8 to 74] | 71.7 [71 to 73] | 71.7 [2 to 73] | 72.0 [48 to 72]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 10 Hours Postdose (AUC0-10) for Metabolite AGI-16903 After a Single Dose of Enasidenib on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3).
  AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 3 | 5 | 3
h*ng/mL | 518.6 (64.5) | 233.3 (30.6) | 1358.2 (46.5) | 965.2 (67.8)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Postdose (AUC0-72) for AGI-16903 After a Single Dose of Enasidenib on Day -3
Description: The first 3 to 5 participants enrolled in each cohort in the dose escalation phase received a single dose of enasidenib three days prior to starting the 28-day dosing regimen (Day -3).
  AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 72 hours post-dose (AUC0-72) was calculated using the linear trapezoidal rule.
Time Frame: Day -3, pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 24, 48, and 72 hours post-dose.
Population: Participants who received 1 dose of enasidenib on Day -3 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 2 | 1 | 4 | 3
h*ng/mL | 7556.4 (42.9) | 7294.2 (99999) | 13752.5 (57.8) | 12519.5 (74.7)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 10 Hours Postdose (AUC0-10) for Enasidenib After Multiple Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3
h*ng/mL | 106522.9 (46.7) | 161862.9 (1.4) | 154248.7 (33.3) | 221865.0 (10.1)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Enasidenib After Multiple Doses
Description: Plasma enasidenib was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 4 | 3
ng/mL | 10717.9 (54.1) | 14945.4 (40.4) | 19401.1 (39.9) | 29316.3 (7.1)

14. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Enasidenib After Multiple Doses
Description: as for outcome 13
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 4 | 3
hours | 8.0 [6 to 10] | 5.9 [1 to 10] | 2.0 [1 to 2] | 2.2 [2 to 8]

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 10 Hours Postdose (AUC0-10) for Metabolite AGI-16903 After Multiple Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
  Area under the plasma concentration-time curve from time 0 to 10 hours post-dose (AUC0-10) was calculated using the linear trapezoidal rule.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 2 | 3 | 3
h*ng/mL | 9074.5 (53.6) | 13914.2 (13.2) | 19865.8 (36.8) | 23007.5 (34.8)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metabolite AGI-16903 After Multiple Doses of Enasidenib
Description: AGI-16903 is a primary metabolite of enasidenib. Plasma AGI-16903 was measured using validated liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 4 | 3
ng/mL | 1093.7 (59.5) | 1435.7 (29.9) | 2101.1 (56.7) | 2837.0 (31.6)

17. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Metabolite AGI-16903 After Multiple Doses of Enasidenib
Description: as for outcome 16
Time Frame: Cycle 2 Day 1 at predose and 0.5, 1, 2, 3, 4, 6, 8, and 10 hours post-dose.
Population: Participants who received enasidenib on Cycle 2 Day 1 with sufficient data to determine PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 4 | 3
hours | 8.0 [2 to 10] | 5.9 [1 to 10] | 1.4 [1 to 2] | 2.2 [2 to 8]

18. Secondary Outcome: Percentage of Participants With Solid Tumors (Excluding Glioma) Who Achieved an Objective Response
Description: Response was assessed based on radiographic evaluations according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria for participants with solid tumors without glioma.
  An objective response was defined as the percentage of participants with complete response (CR) or partial response (PR), confirmed no less than 4 weeks after the criteria for response were first met based on RECIST 1.1.
  Complete response: Disappearance of all target and non-target lesions, pathological lymph nodes must have reduction in short axis to < 10 mm, and no new lesions.
  Partial response: Disappearance of all target lesions with persistence of one or more non-target lesion(s) and/or maintenance of tumor marker levels above the normal limits, or, at least a 30% decrease in the size of target lesions and no progression of existing non-target lesions and no new lesions.
Time Frame: Response assessments were performed every 56 days up to the end of treatment; median (minimum, maximum) duration of treatment was 50.0 (34, 112), 51.5 (41, 57), 40.0 (4, 170), and 27.0 (3, 126) days in each treatment group respectively.
Population: Enrolled participants with solid tumors (excluding glioma) who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 1 | 3 | 3 | 3
percentage of participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Glioma Who Achieved an Objective Response
Description: Response was assessed based on modified Response Assessment in Neuro-Oncology (RANO) working group criteria in participants with glioma.
  An objective response is defined as the percentage of participants with a CR or PR, confirmed no less than 4 weeks based on the modified RANO) criteria.
  CR: Complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks, stable or improved non-enhancing (T2/FLAIR) lesions, no new lesions, participants must be off corticosteroids (or on physiologic replacement doses only), and clinically stable or improved.
  PR: At least 50% decrease compared to Baseline in the size of all measurable enhancing lesions sustained for at least 4 weeks, no progression of non-measurable disease or any new lesions, stable of lower dose of corticosteroids than Baseline dose, and stable or improved non-enhancing (T2/FLAIR) lesions.
Time Frame: as for outcome 18
Population: Enrolled participants with glioma who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 1 | 0 | 4 | 1
percentage of participants | 0 |  | 0 | 0

20. Secondary Outcome: Percentage of Participants With AITL Who Achieved an Objective Response
Description: Response assessments for participants with AITL were based on the revised International Working Group (IWG) Response criteria for Malignant Lymphoma. Overall response was defined as the percentage of participants who achieved a CR or PR based on IWG criteria.
  CR: Disappearance of all evidence of disease, including nodal masses, extra nodal masses, and bone marrow.
  PR: Regression of measurable disease and no new sites (≥ 50% decrease in size from Baseline of all index lesions (both nodal and extranodal lesions), no obvious increase in non-index lesions/disease, fludeoxyglucose (FDG)-avid or positron emission tomography (PET) positive prior to therapy; one or more PET positive at previously involved site, variably FDG-avid or PET negative; regression on computed tomography (CT), no increase in size of liver or spleen).
Time Frame: as for outcome 18
Population: Enrolled participants with AITL who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 1 | 1 | 0 | 3
percentage of participants | 0 | 0 |  | 0

21. Other Pre Specified Outcome: Maximum Increase From Baseline in Corrected QT Interval Based on Fridericia's Formula (QTcF) by Category
Description: QT interval was measured by electrocardiogram throughout the study. The maximum increase in QTcF from Baseline observed across all assessments is reported according to the following categories: increase ≤ 30 milliseconds (ms), increase > 30 to ≤ 60 ms, and increase > 60 ms.
Time Frame: Baseline, Cycle 1 Days 1, 8, 15, and 22, Cycle 2 Days 1 and 15 and Day 1 of every cycle thereafter.
Population: Enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Enasidenb 400 mg: Participants received enasidenib 400 mg tablets QD on Days 1 to 28 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenb 400 mg | Enasidenib 650 mg
Number analyzed (Participants) | 3 | 4 | 6 | 7
Participants
  QTcF Increased from Baseline ≤ 30 ms | 3 | 1 | 5 | 5
  QTcF Increased from Baseline > 30 to ≤ 60 ms | 0 | 3 | 0 | 0
  QTcF Increased from Baseline > 60 ms | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 1 | 0
  no QTcF Increase from Baseline | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 28 days after last dose; median (minimum, maximum) duration of exposure was 66 (8, 197) days across all cohorts.
Arm/Group | Enasidenib 100 mg | Enasidenib 200 mg | Enasidenib 400 mg | Enasidenib 650 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4 | 1/7 | 2/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 3/7 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enasidenib 100 mg (N=3) | Enasidenib 200 mg (N=4) | Enasidenib 400 mg (N=7) | Enasidenib 650 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enasidenib 100 mg (N=3) | Enasidenib 200 mg (N=4) | Enasidenib 400 mg (N=7) | Enasidenib 650 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 3 (4) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (7) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (7) | 4 (4)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (4) | 4 (6) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 2 (11) | 3 (4)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Lipase decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 1 (1) | 1 (2) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was to be conducted in 2 parts: a dose-escalation and an expansion phase. Enrollment was closed after entry into Cohort 4 to focus resources on the development of other pipeline IDH inhibitors in other tumors; there were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.